CLINICAL TRIAL: NCT02542800
Title: ETUDE D'IMAGERIE PAR RESONANCE MAGNETIQUE FONCTIONNELLE CHEZ LE SUJET SAIN DES RELATIONS ENTRE MEMOIRE COLLECTIVE ET INDIVIDUELLE
Brief Title: The Influence of Collective Schemas on Individual Memory (MULTIBRAIN_2)
Acronym: MULTIBRAIN_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: La Région Basse-Normandie (Other); Université de Caen Normandie (Other); University Hospital, Caen (Other); Ecole Pratique des Hautes Etudes (Other); Equipement d'Excellence Matrice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C14-30; 2014-A00650-47 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2017-10

CONDITIONS: Episodic Memory
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy participants (Experimental)
  Interventions: Behavioral: Episodic memory task; Device: fMRI

INTERVENTIONS:
Behavioral: Episodic memory task
Device: fMRI

SUMMARY:
Schemas describe mental structures storing recurrent and organized pattern of information. Schemas may have a strong influence on the process of storing and retrieving new information into memory. Previous approaches in the cognitive neuroscience of memory have entirely focused on the individual dimension of preexisting schemas. In the real world though, much of the researchers' experiences and knowledge are collective or shared. Such social-cultural frameworks stored in collective memory may also reshape and reconfigure the construction of individual memories. Attempting to ascertain the influence of collective schema on the neural substrates of individual memories using cutting-edge brain imaging methods represents the challenge that MULTIBRAIN2 seeks to tackle. To achieve this goal, the researchers will record brain activity during MRI scanning sessions in a group of 24 participants while they are performing an encoding followed by episodic memory retrieval tasks on pictures of the World War II Memorial of Caen. This study will seek to identify brain areas of the prefrontal cortex encoding the organization of knowledge in collective memory using multivariate analyses of brain activity patterns, and then to understand how such regions might modulate the recruitment of the hippocampus during episodic memory retrieval using analyses of effective connectivity. The organization of knowledge in collective memory is measured in parallel through 1) the analysis of French social memory of World War II using a corpus of thousand of television and radio shows from the National Institute of Audiovisual, and 2) an internet task measuring the organization of shared individual knowledge about World War II. Once collected, these data will help us to understand how collective schemas may shape the organization of individual memories.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between 20 and 38 years old
* Affiliated to the French national health care system
* French native speaker
* Having not visited the Memorial of Caen for the past four years
* Right-handed
* At least 2 years of education after graduating from high school
* Body mass < 30kg/m2
* Signed written consent form

Exclusion Criteria:

* Pregnancy or intent to get pregnant
* Person deprived of their liberty
* Person hospitalized without consent
* Minor
* Protected adults or people unable to give informed consent
* Person subjected to an exclusion period related to another protocol
* History of neurological or psychiatric disorders or existence of traumatic brain injury with loss of consciousness for more than one hour
* History of cancer with the last 5 years, excluding squamous cell carcinomas
* Alcoholism, antecedents of chronic alcoholism or drugs abuse
* Severe psychiatric disorders (according to DSM V diagnostic criteria) or psychological troubles which could affect participant's judgment
* Use of medication that may interfere with cognitive or cerebral functioning
* Presence of visual or hearing troubles that may compromise participant's ability to participate in the study
* MRI Contraindications

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) response as measured with fMRI | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Viader, PUPH, Principal Investigator — University Hospital, Caen
Locations (1):
- GIP Cyceron, Caen, France

REFERENCES:
- [Background] Gagnepain P, Vallee T, Heiden S, Decorde M, Gauvain JL, Laurent A, Klein-Peschanski C, Viader F, Peschanski D, Eustache F. Collective memory shapes the organization of individual memories in the medial prefrontal cortex. Nat Hum Behav. 2020 Feb;4(2):189-200. doi: 10.1038/s41562-019-0779-z. Epub 2019 Dec 16. PMID 31844272